CLINICAL TRIAL: NCT04110964
Title: Evaluation of Safety and Tolerability of Libella Gene Therapy (LGT) for Critical Limb Ischemia: AAV- hTERT
Brief Title: Evaluation of Safety and Tolerability of Libella Gene Therapy for Critical Limb Ischemia: AAV- hTERT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Libella Gene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LibellaCO-01
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Critical Limb Ischemia
Keywords: Telomeres; Telomerase; Critical limb ischemia; PAD; AAV; Gene therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- subjects treated with LGT (Experimental): Subjects will be treated with a single IV dose of LGT (AAV-hTERT)
  Interventions: Drug: AAV-hTERT

INTERVENTIONS:
Drug: AAV-hTERT — subjects will receive a single LGT (AAV-hTERT) treatment via IV administration
  Other Names: LGT

SUMMARY:
Using gene therapy to express active telomerase (hTERT) in human cells has the potential to treat many diseases related to aging, including critical limb ischemia (CLI).

This study will entail treating subjects with hTERT delivered via transduction using AAV. The goal is to extend the telomeres to prevent, delay, or even reverse the development of the pathology of CLI. It is expected to have a direct consequence on function and quality of life in patients with Peripheral artery disease (PAD); in this case a subgroup of patients with CLI, the worst presentation of PAD.

DETAILED DESCRIPTION:
Patients diagnosed with CLI who meet with the inclusion - exclusion criteria, will be treated with a single dose of LGT delivered intravascularly (IV).

Baseline will be performed within 8 weeks of beginning the treatment regimen. The treatment regimen will begin with IV delivery of AAV-hTERT, defined as "Day 0." Safety and efficacy analyses will be conducted at Weeks 1, 4, 13, 26, 39, and 52 post-treatment.

Study objectives

Primary: Safety and Tolerability

1. Investigate the safety and tolerability of AAV-hTERT by intravenous (IV) administration.

Secondary: Provisional Efficacy

1. Investigate LGT's ability to deliver hTERT to human cells and lengthen telomeres.
2. Investigate the effects of lengthening telomeres on CLI.
3. Investigate other benefits provided by lengthening telomeres.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 45 years or older.
2. Clinical diagnosis of CLI.
3. Subjects, or their authorized representatives, must be adequately informed and understand the nature and risks of the study and must be able to provide a signature and date in the Informed Consent Form (ICF).
4. Women must undergo a negative serum pregnancy test at the screening assessment.
5. Subjects, or their representatives, must be able to communicate effectively with the study staff.
6. Subjects, or their authorized representatives, must certify that they are able and willing to follow all protocol requirements and study restrictions.

Exclusion Criteria:

1. Subjects who have a history of allergy, hypersensitivity, or intolerance to any medications, components, or excipients of the investigational product, which cannot be resolved by the staff conducting the study.
2. Female subjects who are pregnant, expected to become pregnant, or lactating/nursing.
3. Subjects who are sexually active and who are unwilling or unable to use a method of effective contraception (e.g., hormonal and/or barrier) during their participation in the study.
4. Subjects who are intolerant of, or do not wish to receive IV injections.
5. Subjects who are currently alcoholics and/or use psychoactive substances.
6. Subjects who cannot tolerate venipuncture and/or venous access.
7. Subjects who have donated or had a significant loss of whole blood (480 ml or more) within 30 days, or donated plasma or platelets within 14 days prior to screening.
8. Subjects who have received blood or blood products within 30 days prior to screening.
9. Subjects who have been treated with another research product 30 days prior to the screening assessment, or plan to participate in another clinical trial, while in this study if in the opinion of the principal investigator, may place the subject at risk due to participation in the study, or may influence the results of the study or the subject's ability to complete the study. If more than 30 days have passed since participation in another clinical trial, the study staff must ensure that the subject has recovered from any adverse event (AE) associated with the research product used.
10. Subjects who have a history or evidence of active infection or febrile illness within 7 days prior to the screening assessment.

Subjects who have a history of any other clinically significant disease or disorder that, in the opinion of the principal investigator, may place the subject at risk due to participation in the study, or may influence the results of the study or the subject's ability to complete the study.

-

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 months
  Incidence of serious adverse events and adverse events throughout the study

SECONDARY OUTCOMES:
hTERT expression and telomerase activity | 12 months
  Change from baseline of the telomere length

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Ulloa, MD, Principal Investigator — IPS Arcaslud SAS
Locations (1):
- IPS Arcasalud SAS, Zipaquirá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No